CLINICAL TRIAL: NCT04102995
Title: An Exploratory Phase II, Randomised, Double-blind, Placebo-controlled, Parallel-group Study Investigating the Efficacy and Safety of Sepranolone in Women With Menstrual Migraine
Brief Title: A Study Investigating the Efficacy and Safety of Sepranolone in Women With Menstrual Migraine
Acronym: APH204
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asarina Pharma (Industry)
Collaborators: Aurevia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APH204
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Menstrual Migraine
MeSH Terms: interventions — Pregnanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sepranolone (UC1010) low dose (Experimental): Subcutaneous injection every 48 hours during the luteal phase during three menstrual cycles in women with menstrual migraine
  Interventions: Drug: Sepranolone injection low dose
- Sepranolone (UC1010) high dose (Experimental): Subcutaneous injection every 48 hours during the luteal phase during three menstrual cycles in women with menstrual migraine
  Interventions: Drug: Sepranolone injection high dose
- Placebo (Placebo Comparator): Subcutaneous injection every 48 hours during the luteal phase during three menstrual cycles in women with menstrual migraine
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Sepranolone injection low dose — Subcutaneous (SC) administration
  Other Names: UC1010
  Arms: Sepranolone (UC1010) low dose
Drug: Sepranolone injection high dose — Subcutaneous (SC) administration
  Other Names: UC1010
  Arms: Sepranolone (UC1010) high dose
Drug: Placebo injection — Subcutaneous (SC) administration
  Arms: Placebo

SUMMARY:
The objective of this phase 2 Proof.of Concept study is to evaluate the efficacy and safety of Sepranolone (UC1010) in preventing menstrual migraine attacks in adult women with migraine occurring between Day -2 and Day 5 of the menstrual cycle. Patients will be taking Sepranolone or Placebo (blinded to patient and study doctor) during the two week preceding the menstruation for three menstrual cycles. Effect (change from baseline) will be assessed by comparison of symptoms recorded daily by the patients using an electronic diary using validated scales for assessment of menstual migraine symptoms.

Sepranolone is identical to an endogenous steroid.

DETAILED DESCRIPTION:
The objective of this phase 2 Proof-of-Concept study is to evaluate the effect and safety of two doses of Sepranolone (UC1010) in preventing menstrual migraine attacks in adult women with migraine occurring between Day -2 and Day 5 of the menstrual cycle in comparison to placebo. Study treatment will be self-administrated as subcutaneous injections during the luteal phase of three consecutive menstrual cycles. Effect will be assessed by comparison of symptoms recorded daily by the patients using an electronic migraine diary and a validated rating scale for assessment the physical and functional impact of menstrual migraine symptoms (MPFID). Preceding the treatment period, the diagnosis of Menstrual Migraine will be established by verifying menstrual migraine in at least two out of three menstrual cycles of daily symptom ratings by the patients. This period will also constitute the baseline data. The effect of study medication will be assessed as the change in symptoms from baseline to during treatment. The reduction in average number of menstrual migraine days per menstrual cycle during the treatment period cycles vs. the three menstrual cycles of baseline will constitute the primary endpoint.

The study will also include a follow-up (no treatment) cycle before patients final visit.

The study is conducted in three European countries (Sweden, Finland and Denmark) and will randomize 84 patients.

ELIGIBILITY:
Inclusion Criteria:

* have Menstrual Migraine according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) verified in three menstrual cycles
* have a regular menstrual cycle of 24-35 days cycle,
* use double barrier contraception, intrauterine device (IUD), be truly sexually abstinent, or subject or her partner has been surgically sterilized,

Exclusion Criteria:

* More than 10 headache days per month on average during screening phase
* steroid hormonal treatment during previous three months
* ongoing treatment with antiepileptic drugs or benzodiazepines
* significant medical or psychiatric condition
* be pregnant or plan a pregnancy within the study period

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Change in number of menstrual migraine days | Through study completion, an average of 6 months
  Change from baseline in the average number of menstrual migraine days during three consecutive menstrual cycles

CONTACTS AND LOCATIONS:
Locations (7):
- Finland (3):
  - Suomen Terveystalo Plc, Helsinki
  - Suomen Terveystalo Plc, Tampere
  - Suomen Terveystalo Plc, Turku
- Sweden (4):
  - ProbarE i Lund, Lund, Skåne County
  - CTC Clinical Trial Center, Gothenburg
  - Karolinska Trial Alliance, Stockholm
  - CTC Clinical Trial Consultants, Uppsala

IPD SHARING:
Plan to Share IPD: No